CLINICAL TRIAL: NCT00253669
Title: Pilot Study of Thrombophilic States in Newly Diagnosed Patients With High-Grade Gliomas
Brief Title: Risk Factors for Developing a Blood Clot in Patients Who Are Undergoing Cancer Treatment for Newly Diagnosed Gliomas
Status: Completed | Type: Observational
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH); North American Brain Tumor Consortium (Other)
Responsible Party: Sponsor
Other Study IDs: NABTT-0307; U01CA062475 (NIH); CDR0000441111; JHOC-NABTT-0307
Record Dates: First submitted 2005-11-11; First posted 2005-11-15 (Estimated); Last update posted 2018-06-28 (Actual); Status verified 2018-06

CONDITIONS: Brain and Central Nervous System Tumors; Thromboembolism
Keywords: thromboembolism; adult anaplastic astrocytoma; adult anaplastic oligodendroglioma; adult glioblastoma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Thromboembolism; Astrocytoma; Oligodendroglioma; Glioblastoma; Gliosarcoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

INTERVENTIONS:
Other: laboratory biomarker analysis
Other: physiologic testing
Procedure: management of therapy complications

SUMMARY:
RATIONALE: Patients with gliomas may be at risk for developing blood clots. Learning about the risk factors for developing blood clots may help doctors plan better treatment for gliomas.

PURPOSE: This clinical trial is studying risk factors for developing blood clots in patients who are undergoing cancer treatment for newly diagnosed gliomas.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the overall hazard rate of first venous thromboembolism per person-year of follow-up in patients undergoing antineoplastic therapy for newly diagnosed high-grade gliomas.
* Correlate ABO blood type with incidence of venous thromboembolism in these patients.
* Correlate factor VIII level with incidence of venous thromboembolism in these patients.

Secondary

* Determine the overall and individual incidence rate of thromboembolism in these patients.
* Correlate clinical variables, such as type of antineoplastic treatments, Karnofsky performance status, and type of tumor, with incidence of venous thromboembolism in these patients.
* Correlate demographic factors, such as age, with incidence of venous thromboembolism in these patients.

OUTLINE: This is a pilot, multicenter study.

Patients undergo blood collection for blood typing (if not already obtained) and factor VIII and C-reactive protein levels at baseline. Patients are followed to obtain information on their Karnofsky performance status, treatment they receive for their brain tumor, and occurrence of any thrombotic events (e.g., pulmonary embolism or deep-vein thrombosis). Patients are followed every 28 days until the development of thrombotic events, after which they are followed every 2 months for survival.

PROJECTED ACCRUAL: A total of 107 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed newly diagnosed malignant brain tumor

  * Supratentorial grade III or IV astrocytoma of 1 of the following types:

    * Anaplastic astrocytoma
    * Anaplastic oligodendroglioma
    * Glioblastoma multiforme
* No prior thrombotic event

PATIENT CHARACTERISTICS:

Performance status

* Karnofsky 60-100%

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior immunotherapy or biologic agents, including immunotoxins, immunoconjugates, antisense therapy, peptide-receptor antagonists, interferons, interleukins, tumor-infiltrating lymphocytes, lymphocyte-activated killer cells, or gene therapy, for the brain tumor

Chemotherapy

* No prior chemotherapy for the brain tumor except polifeprosan 20 with carmustine implant (Gliadel wafer)

Endocrine therapy

* No prior hormonal therapy for the brain tumor except glucocorticoids

Radiotherapy

* No prior radiotherapy for the brain tumor
* No prior cranial irradiation

Other

* No concurrent chronic anticoagulation therapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: outpatient clinic
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2005-04; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Thrombosis-free survival as assessed by objectively documented deep vein thrombosis or pulmonary embolism | until dvt or death

SECONDARY OUTCOMES:
ABO blood group association with venous thromboembolism (VTE) factor VIII activity and VTE as assessed by laboratory test result at study entry | on study

CONTACTS AND LOCATIONS:
Overall Officials: Michael B. Streiff, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins; Stuart A. Grossman, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins; Larry Kleinberg, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (9):
- United States (9):
  - Lurleen Wallace Comprehensive Cancer at University of Alabama - Birmingham, Birmingham, Alabama
  - H. Lee Moffitt Cancer Center and Research Institute at University of South Florida, Tampa, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania